CLINICAL TRIAL: NCT00381030
Title: Effects of Inpatient Initiation of Carvedilol and Nurse Management on Health Outcomes in Vulnerable Heart Failure Patients (ECHO Study): a Randomized Trial
Brief Title: Effects of Carvedilol on Health Outcomes in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKF105517/379
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2006-09-27 (Estimated); Status verified 2006-09

CONDITIONS: Heart Failure, Congestive
Keywords: beta-Adrenergic Blockers; Disease Management
MeSH Terms: conditions — Heart Failure | interventions — Carvedilol

INTERVENTIONS:
Drug: carvedilol plus nurse management

SUMMARY:
The purpose of our study was to determine if a strategy of starting a heart medication (Beta-blocker) before patients leave the hospital and then being seen by a nurse manager would reduce subsequent hospitalizations compared to usual care.

Hypothesis: A nurse-directed heart failure management program with inpatient initiation of beta blockers will improve health outcomes in a vulnerable, predominantly Hispanic and African American population.

DETAILED DESCRIPTION:
Heart failure is a leading cause of death and hospitalization in the US. Designing practical approaches to improving heart failure care is therefore a national health priority. One retrospective study suggested that patients taking beta-blockers while hospitalized for heart failure had a lower risk of rehospitalization at 6-months. One prospective study suggested that starting beta blockers among hospitalized heart failure patients is safe and improves compliance. However, improved outcomes of this approach have not been prospectively demonstrated.

Comparison: Inpatient initiation of the beta-blocker carvedilol coupled with outpatient follow-up with a nurse manager was compared to usual care by internists and cardiologists.

ELIGIBILITY:
Inclusion Criteria:

* primary hospitalization with heart failure and LVEF < 40%
* patient informed consent has been obtained
* absence of pulmonary congestion
* age > 18 years

Exclusion Criteria:

* End-stage renal or hepatic disease
* Acute myocardial infarction as primary diagnosis during index hospitalization
* Life-expectancy < 6-months
* Contraindication to beta blocker use
* Current beta-blocker therapy
* Planned bypass or valve surgery during index hospitalization

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2002-10; Study Completion 2005-03

PRIMARY OUTCOMES:
Primary outcome: heart failure hospitalizations, time to death or hospitalization

SECONDARY OUTCOMES:
left ventricular ejection fraction and volume in systole and diastole
beta-blocker utilization/adherence
new york heart association functional class

CONTACTS AND LOCATIONS:
Overall Officials: Mori J Krantz, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Krantz MJ, Havranek EP, Haynes DK, Smith I, Bucher-Bartelson B, Long CS. Inpatient initiation of beta-blockade plus nurse management in vulnerable heart failure patients: a randomized study. J Card Fail. 2008 May;14(4):303-9. doi: 10.1016/j.cardfail.2007.12.008. PMID 18474343